CLINICAL TRIAL: NCT01107418
Title: A Phase I, Randomized, Open-label, Multi-center, Multiple Dose Study to Investigate the Pharmacokinetics and Pharmacodynamics of RO5185426 Administered as 240 mg Tablets to Previously Treated BRAF V600E Positive Metastatic Melanoma Patients
Brief Title: A Pharmacokinetic/Pharmacodynamic Study of RO5185426 in Previously Treated Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP25163
Record Dates: First submitted 2010-04-12; First posted 2010-04-21 (Estimated); Results first posted 2015-08-26 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-07

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: RO5185426
- 2 (Experimental)
  Interventions: Drug: RO5185426
- 3 (Experimental)
  Interventions: Drug: RO5185426
- 4 (Experimental)
  Interventions: Drug: RO5185426

INTERVENTIONS:
Drug: RO5185426 — dosage b) orally twice daily, days 1-15 (morning dose)
  Arms: 2
Drug: RO5185426 — dosage c) orally twice daily, days 1-15 (morning dose)
  Arms: 3
Drug: RO5185426 — dosage d) orally twice daily, days 1-15 (morning dose)
  Arms: 4
Drug: RO5185426 — 960 mg orally twice daily, from day 22 onward
Drug: RO5185426 — dosage a) orally twice daily, days 1-15 (morning dose)
  Arms: 1

SUMMARY:
This open-label study will assess the pharmacokinetics, efficacy and safety of RO5185426 administered as 240mg tablets in previously treated patients with metastatic melanoma. Patients will be randomized to receive one of four dose-levels of RO5185426 [RG7204; PLEXXIKON; PLX4032] orally twice daily on days 1 to 15 (morning dose). Starting on day 22, treatment with RO5185426 may be resumed at a dose of 960 mg twice daily and continued until disease progression. Target sample size is <100 patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/=18 years of age
* histologically confirmed metastatic melanoma, stage IIIc or IV (AJCC)
* failure of at least one prior standard of care regimen
* positive for BRAF V600E mutation (by Roche CoDx BRAF mutation assay)
* ECOG performance status 0 or 1
* adequate hematologic, renal and liver function

Exclusion Criteria:

* active CNS lesions on CT/MRI within 28 days prior to enrollment
* history of spinal cord compression o carcinomatous meningitis
* anticipated or ongoing anti-cancer therapies other than those administered in this study
* previous treatment with BRAF inhibitor (sorafenib allowed) or MEK inhibitor
* severe cardiovascular disease within 6 months prior to study
* previous malignancy within the past 5 years except for basal or squamous cell carcinoma of the skin, melanoma in-situ and carcinoma in-situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- United States (11):
  - La Jolla, California
  - San Francisco, California
  - Stanford, California
  - New Haven, Connecticut
  - Chicago, Illinois
  - Park Ridge, Illinois
  - Sioux City, Iowa
  - Omaha, Nebraska
  - Columbus, Ohio
  - East Providence, Rhode Island
  - Charlottesville, Virginia
- Australia (2):
  - Adelaide, South Australia
  - Melbourne, Victoria

REFERENCES:
- [Derived] Frederick DT, Salas Fragomeni RA, Schalck A, Ferreiro-Neira I, Hoff T, Cooper ZA, Haq R, Panka DJ, Kwong LN, Davies MA, Cusack JC, Flaherty KT, Fisher DE, Mier JW, Wargo JA, Sullivan RJ. Clinical profiling of BCL-2 family members in the setting of BRAF inhibition offers a rationale for targeting de novo resistance using BH3 mimetics. PLoS One. 2014 Jul 1;9(7):e101286. doi: 10.1371/journal.pone.0101286. eCollection 2014. PMID 24983357
- [Derived] Lacouture ME, Duvic M, Hauschild A, Prieto VG, Robert C, Schadendorf D, Kim CC, McCormack CJ, Myskowski PL, Spleiss O, Trunzer K, Su F, Nelson B, Nolop KB, Grippo JF, Lee RJ, Klimek MJ, Troy JL, Joe AK. Analysis of dermatologic events in vemurafenib-treated patients with melanoma. Oncologist. 2013;18(3):314-22. doi: 10.1634/theoncologist.2012-0333. Epub 2013 Mar 1. PMID 23457002

RESULTS

PARTICIPANT FLOW:
Groups:
- Vemurafenib - All Cohorts: Participants received vemurafenib (RO5185426) film-coated tablets, orally, twice daily at doses of 240, 480, 720, or 960 milligrams (mg) on Days 1 to 15 (a single morning dose was administered on Day 15). Starting at Day 22, participants received vemurafenib 960 mg film-coated tablets orally twice daily in 21-day cycles until the development of progressive disease, unacceptable toxicity, consent withdrawal, or any other criteria for removal.
Period: Overall Study
Arm/Group | Vemurafenib - All Cohorts
Started | 52
Completed | 0
Not Completed | 52
Not completed — Disease Progression | 45
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Study Closing | 1
Not completed — Started Other Therapy | 1
Not completed — Entered Extension Study | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of vemurafenib.
Groups:
- Cohort 1 - Vemurafenib 240 mg: Participants received vemurafenib film-coated tablet, orally, twice daily at a dose of 240 mg on Days 1 to 15 (a single morning dose was administered on Day 15). Starting at Day 22, participants received vemurafenib 960 mg film-coated tablets orally twice daily in 21-day cycles until the development of progressive disease, unacceptable toxicity, consent withdrawal, or any other criteria for removal.
- Cohort 2 - Vemurafenib 480 mg: Participants received vemurafenib film-coated tablets, orally, twice daily at a dose of 480 mg on Days 1 to 15 (a single morning dose was administered on Day 15). Starting at Day 22, participants received vemurafenib 960 mg film-coated tablets orally twice daily in 21-day cycles until the development of progressive disease, unacceptable toxicity, consent withdrawal, or any other criteria for removal.
- Cohort 3 - Vemurafenib 720 mg: Participants received vemurafenib film-coated tablets, orally, twice daily at a dose of 720 mg on Days 1 to 15 (a single morning dose was administered on Day 15). Starting at Day 22, participants received vemurafenib 960 mg film-coated tablets orally twice daily in 21-day cycles until the development of progressive disease, unacceptable toxicity, consent withdrawal, or any other criteria for removal.
- Cohort 4 - Vemurafenib 960 mg: Participants received vemurafenib film-coated tablets, orally, twice daily at a dose of 960 mg on Days 1 to 15 (a single morning dose was administered on Day 15). Starting at Day 22, participants resumed vemurafenib 960 mg film-coated tablets orally twice daily in 21-day cycles until the development of progressive disease, unacceptable toxicity, consent withdrawal, or any other criteria for removal.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Vemurafenib 240 mg | Cohort 2 - Vemurafenib 480 mg | Cohort 3 - Vemurafenib 720 mg | Cohort 4 - Vemurafenib 960 mg | Total
Number analyzed (Participants) | 12 | 12 | 12 | 16 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (15.06) | 46.3 (10.58) | 54.3 (10.70) | 50.5 (11.91) | 50.8 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 6 | 8 | 26
  Male | 7 | 5 | 6 | 8 | 26

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 8 Hours (AUC[0-8h]) of Vemurafenib on Day 1
Time Frame: Pre-dose, 1, 2, 4, 5, 8 hours post-dose on Day 1
Population: Pharmacokinetic (PK) population included all participants who provided essential PK data up to and including the pre-dose PK sample taken on Cycle 1, Day 22, without major protocol violation.
Measure: Mean (Standard Deviation); unit: micrograms*hour/milliliter (mcg*h/mL)
Arm/Group | Cohort 1 - Vemurafenib 240 mg | Cohort 2 - Vemurafenib 480 mg | Cohort 3 - Vemurafenib 720 mg | Cohort 4 - Vemurafenib 960 mg
Number analyzed (Participants) | 12 | 12 | 12 | 16
micrograms*hour/milliliter (mcg*h/mL) | 8.3 (6.13) | 13.8 (7.72) | 21.9 (12.97) | 27.0 (18.87)

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC[0-24h]) of Vemurafenib on Day 1
Time Frame: Pre-dose, 1, 2, 4, 5, 8, 24 hours post-dose on Day 1
Population: PK population. Here, number of participants analyzed signifies participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Cohort 1 - Vemurafenib 240 mg | Cohort 2 - Vemurafenib 480 mg | Cohort 3 - Vemurafenib 720 mg | Cohort 4 - Vemurafenib 960 mg
Number analyzed (Participants) | 11 | 12 | 9 | 16
mcg*h/mL | 40.9 (23.43) | 62.4 (35.71) | 111.6 (34.22) | 130.6 (71.78)

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of Vemurafenib on Day 1
Time Frame: Pre-dose, 1, 2, 4, 5, 8 hours post-dose on Day 1
Population: PK population.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter (mcg/mL)
Arm/Group | Cohort 1 - Vemurafenib 240 mg | Cohort 2 - Vemurafenib 480 mg | Cohort 3 - Vemurafenib 720 mg | Cohort 4 - Vemurafenib 960 mg
Number analyzed (Participants) | 12 | 12 | 12 | 16
micrograms/milliliter (mcg/mL) | 1.9 (1.66) | 2.6 (1.56) | 4.4 (1.98) | 4.8 (3.34)

4. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Vemurafenib on Day 1
Time Frame: Pre-dose, 1, 2, 4, 5, 8 hours post-dose on Day 1
Population: PK population.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 - Vemurafenib 240 mg | Cohort 2 - Vemurafenib 480 mg | Cohort 3 - Vemurafenib 720 mg | Cohort 4 - Vemurafenib 960 mg
Number analyzed (Participants) | 12 | 12 | 12 | 16
hours | 4.0 [1.92 to 8.00] | 4.0 [1.95 to 5.00] | 5.0 [2.00 to 8.08] | 5.0 [2.00 to 8.00]

5. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 8 Hours (AUC[0-8h]) of Vemurafenib on Day 9
Time Frame: Pre-dose, 1, 2, 4, 5, 8 hours post-dose on Day 9
Population: PK population. Here, number of participants analyzed signifies participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Cohort 1 - Vemurafenib 240 mg | Cohort 2 - Vemurafenib 480 mg | Cohort 3 - Vemurafenib 720 mg | Cohort 4 - Vemurafenib 960 mg
Number analyzed (Participants) | 11 | 11 | 9 | 12
mcg*h/mL | 102.1 (41.37) | 180.0 (84.23) | 301.2 (108.67) | 329.0 (108.85)

6. Primary Outcome: Maximum Plasma Concentration (Cmax) of Vemurafenib on Day 9
Time Frame: Pre-dose, 1, 2, 4, 5, 8 hours post-dose on Day 9
Population: PK population. Here, number of participants analyzed signifies participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort 1 - Vemurafenib 240 mg | Cohort 2 - Vemurafenib 480 mg | Cohort 3 - Vemurafenib 720 mg | Cohort 4 - Vemurafenib 960 mg
Number analyzed (Participants) | 11 | 11 | 9 | 12
mcg/mL | 15.4 (5.84) | 28.9 (16.95) | 45.9 (14.44) | 53.2 (19.08)

7. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Vemurafenib on Day 9
Time Frame: Pre-dose, 1, 2, 4, 5, 8 hours post-dose on Day 9
Population: PK population. Here, number of participants analyzed signifies participants evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 - Vemurafenib 240 mg | Cohort 2 - Vemurafenib 480 mg | Cohort 3 - Vemurafenib 720 mg | Cohort 4 - Vemurafenib 960 mg
Number analyzed (Participants) | 11 | 11 | 9 | 12
hours | 2.0 [0.00 to 8.00] | 2.0 [0.00 to 5.08] | 0.0 [0.00 to 8.00] | 1.8 [0.00 to 8.00]

8. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 8 Hours (AUC[0-8h]) of Vemurafenib on Day 15
Time Frame: Pre-dose, 1, 2, 4, 5, 8 hours post-dose on Day 15
Population: PK population. Here, number of participants analyzed signifies participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Cohort 1 - Vemurafenib 240 mg | Cohort 2 - Vemurafenib 480 mg | Cohort 3 - Vemurafenib 720 mg | Cohort 4 - Vemurafenib 960 mg
Number analyzed (Participants) | 10 | 9 | 9 | 11
mcg*h/mL | 117.8 (50.52) | 233.8 (106.93) | 343.3 (151.23) | 392.2 (126.37)

9. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC[0-24h]) of Vemurafenib on Day 15
Time Frame: Pre-dose, 1, 2, 4, 5, 8, 24 hours post-dose on Day 15
Population: PK population. Here, number of participants analyzed signifies participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Cohort 1 - Vemurafenib 240 mg | Cohort 2 - Vemurafenib 480 mg | Cohort 3 - Vemurafenib 720 mg | Cohort 4 - Vemurafenib 960 mg
Number analyzed (Participants) | 10 | 10 | 9 | 11
mcg*h/mL | 317.7 (133.34) | 598.8 (297.44) | 1003.7 (441.36) | 1126.0 (423.01)

10. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 168 Hours (AUC[0-168h]) of Vemurafenib on Day 15
Time Frame: Pre-dose, 1, 2, 4, 5, 8, 24, 28, 72, 76, 168 hours post-dose on Day 15
Population: PK population. Here, number of participants analyzed signifies participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Cohort 1 - Vemurafenib 240 mg | Cohort 2 - Vemurafenib 480 mg | Cohort 3 - Vemurafenib 720 mg | Cohort 4 - Vemurafenib 960 mg
Number analyzed (Participants) | 10 | 8 | 9 | 11
mcg*h/mL | 920.3 (538.35) | 2243.5 (1336.15) | 3127.1 (1789.97) | 3530.3 (1811.43)

11. Primary Outcome: Maximum Plasma Concentration (Cmax) of Vemurafenib on Day 15
Time Frame: Pre-dose, 1, 2, 4, 5, 8, 24, 28, 72, 76, 168 hours post-dose on Day 15
Population: PK population. Here, number of participants analyzed signifies participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort 1 - Vemurafenib 240 mg | Cohort 2 - Vemurafenib 480 mg | Cohort 3 - Vemurafenib 720 mg | Cohort 4 - Vemurafenib 960 mg
Number analyzed (Participants) | 10 | 9 | 9 | 11
mcg/mL | 17.2 (7.43) | 35.4 (17.44) | 52.7 (22.40) | 61.4 (22.76)

12. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Vemurafenib on Day 15
Time Frame: Pre-dose, 1, 2, 4, 5, 8, 24, 28, 72, 76, 168 hours post-dose on Day 15
Population: PK population. Here, number of participants analyzed signifies participants evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 - Vemurafenib 240 mg | Cohort 2 - Vemurafenib 480 mg | Cohort 3 - Vemurafenib 720 mg | Cohort 4 - Vemurafenib 960 mg
Number analyzed (Participants) | 10 | 9 | 9 | 11
hours | 4.0 [0.00 to 8.00] | 2.3 [0.00 to 5.00] | 2.0 [0.00 to 24.17] | 2.0 [0.00 to 24.00]

13. Primary Outcome: Apparent Clearance (CL/F) of Vemurafenib on Day 15
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Time Frame: Pre-dose, 1, 2, 4, 5, 8, 24, 28, 72, 76, 168 hours post-dose on Day 15
Population: PK population. Here, number of participants analyzed signifies participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: liters/hour (L/h)
Arm/Group | Cohort 1 - Vemurafenib 240 mg | Cohort 2 - Vemurafenib 480 mg | Cohort 3 - Vemurafenib 720 mg | Cohort 4 - Vemurafenib 960 mg
Number analyzed (Participants) | 10 | 8 | 9 | 11
liters/hour (L/h) | 0.3 (0.13) | 0.8 (1.45) | 0.4 (0.28) | 0.3 (0.19)

14. Primary Outcome: Terminal Elimination Half-Life (t1/2) of Vemurafenib on Day 15
Description: Time measured for vemurafenib plasma concentrations to decrease by one-half (t1/2) was calculated as 0.693 divided by apparent first-order terminal elimination rate constant (0.693/kel).
Time Frame: Pre-dose, 1, 2, 4, 5, 8, 24, 28, 72, 76, 168 hours post-dose on Day 15
Population: PK population. Here, number of participants analyzed signifies participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Cohort 1 - Vemurafenib 240 mg: Participants received vemurafenib film-coated tablets, orally, twice daily at a dose of 240 mg on Days 1 to 15 (a single morning dose was administered on Day 15). Starting at Day 22, participants received vemurafenib 960 mg film coated tablet twice daily orally in 21-day cycles until the development of progressive disease, unacceptable toxicity, consent withdrawal, or any other criteria for removal.
- Cohort 2 - Vemurafenib 480 mg: Participants received vemurafenib film-coated tablets, orally, twice daily at a dose of 480 mg on Days 1 to 15 (a single morning dose was administered on Day 15). Starting at Day 22, participants received vemurafenib 960 mg film coated tablet twice daily orally in 21-day cycles until the development of progressive disease, unacceptable toxicity, consent withdrawal, or any other criteria for removal.
- Cohort 3 - Vemurafenib 720 mg: Participants received vemurafenib film-coated tablets, orally, twice daily at a dose of 720 mg on Days 1 to 15 (a single morning dose was administered on Day 15). Starting at Day 22, participants received vemurafenib 960 mg film coated tablet twice daily orally in 21-day cycles until the development of progressive disease, unacceptable toxicity, consent withdrawal, or any other criteria for removal.
- Cohort 4 - Vemurafenib 960 mg: Participants received vemurafenib film-coated tablets, orally, twice daily at a dose of 960 mg on Days 1 to 15 (a single morning dose was administered on Day 15). Starting at Day 22, participants received vemurafenib 960 mg film coated tablet twice daily orally in 21-day cycles until the development of progressive disease, unacceptable toxicity, consent withdrawal, or any other criteria for removal.
Arm/Group | Cohort 1 - Vemurafenib 240 mg | Cohort 2 - Vemurafenib 480 mg | Cohort 3 - Vemurafenib 720 mg | Cohort 4 - Vemurafenib 960 mg
Number analyzed (Participants) | 10 | 10 | 9 | 11
hours | 31.5 (19.05) | 38.4 (24.18) | 34.9 (19.48) | 34.1 (19.66)

15. Secondary Outcome: Percentage of Participants With a Confirmed Best Overall Response of Complete Response (CR) or Partial Response (PR)
Description: Confirmed best overall response was defined as having best objective response as CR or PR, as assessed by investigator and confirmed at least 28 days after initial response. Tumor response was assessed according to the Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1). CR was defined as the disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) were required to demonstrate a reduction to normal (short axis less than [<] 10 millimeters [mm]). PR was defined as a 30 percent (%) decrease in the sum of the diameters of the target lesions taking as a reference the baseline sum diameter. Percentage of participants with best overall response of confirmed CR or PR are reported.
Time Frame: Up to approximately 3 years (assessed at Cycle 1 Day 1, Cycle 3 Day 1, Cycle 5 Day 1, thereafter every 2 cycles and then every 4 cycles after Cycle 13)
Population: Efficacy population: all enrolled participants who received at least one dose of vemurafenib, had measurable target lesions at baseline based on RECIST 1.1 criteria, had no major protocol violations of inclusion/exclusion criteria, and had no other violations affecting efficacy assessments.
Measure: Number; unit: percentage of participants
Groups:
- Vemurafenib - All Cohorts: Participants received vemurafenib film-coated tablets, orally, twice daily at doses of 240, 480, 720, or 960 mg on Days 1 to 15 (a single morning dose was administered on Day 15). Starting at Day 22, participants received vemurafenib 960 mg film-coated tablets orally twice daily in 21-day cycles until the development of progressive disease, unacceptable toxicity, consent withdrawal, or any other criteria for removal.
Arm/Group | Vemurafenib - All Cohorts
Number analyzed (Participants) | 49
percentage of participants | 49

16. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time, in months, from the date of the first study drug administration to the date of death, regardless of the cause of death.
Time Frame: as for outcome 15
Population: Data for this outcome measure was not collected as the outcome was removed as per changes in planned analysis (protocol amendment).
Arm/Group | Vemurafenib - All Cohorts
Number analyzed (Participants) | 0

17. Primary Outcome: Accumulation Ratio of Vemurafenib on Day 15
Description: Accumulation ratio was calculated as, AUC(0-8) on Day 15 divided by AUC(0-8) on Day 1.
Time Frame: Pre-dose, 1, 2, 4, 5, 8 hours post-dose on Day 1 and 15
Population: PK population. Here, number of participants analyzed signifies participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 1 - Vemurafenib 240 mg | Cohort 2 - Vemurafenib 480 mg | Cohort 3 - Vemurafenib 720 mg | Cohort 4 - Vemurafenib 960 mg
Number analyzed (Participants) | 10 | 9 | 9 | 11
ratio | 24.9 (29.4) | 23.3 (16.0) | 18.8 (12.4) | 23.2 (16.5)

ADVERSE EVENTS:
Time Frame: Up to approximately 3 years
Arm/Group | Cohort 1 - Vemurafenib 240 mg | Cohort 2 - Vemurafenib 480 mg | Cohort 3 - Vemurafenib 720 mg | Cohort 4 - Vemurafenib 960 mg
Serious Adverse Events (participants affected / at risk) | 3/12 | 3/12 | 8/12 | 7/16
Other Adverse Events (participants affected / at risk) | 12/12 | 12/12 | 12/12 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Vemurafenib 240 mg (N=12) | Cohort 2 - Vemurafenib 480 mg (N=12) | Cohort 3 - Vemurafenib 720 mg (N=12) | Cohort 4 - Vemurafenib 960 mg (N=16)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2 | 2
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 2
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Shock (Vascular disorders) | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Vemurafenib 240 mg (N=12) | Cohort 2 - Vemurafenib 480 mg (N=12) | Cohort 3 - Vemurafenib 720 mg (N=12) | Cohort 4 - Vemurafenib 960 mg (N=16)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 4
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Keratosis follicular (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Porokeratosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Cushingoid (Endocrine disorders) | 0 | 1 | 0 | 0
Binocular eye movement disorder (Eye disorders) | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 2
Diplopia (Eye disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 1 | 0
Episcleritis (Eye disorders) | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 1 | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 1
Eyelid irritation (Eye disorders) | 0 | 0 | 0 | 1
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 0
Ocular discomfort (Eye disorders) | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 1
Pupils unequal (Eye disorders) | 0 | 1 | 0 | 0
Retinal disorder (Eye disorders) | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 6 | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 5 | 5 | 6
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 5 | 6 | 7
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Salivary gland calculus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Salivary gland mass (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 3 | 2 | 5
Asthenia (General disorders) | 1 | 0 | 3 | 1
Axillary pain (General disorders) | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 1 | 1
Chills (General disorders) | 0 | 1 | 2 | 2
Cyst (General disorders) | 1 | 1 | 0 | 2
Early satiety (General disorders) | 0 | 0 | 1 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 1
Fatigue (General disorders) | 10 | 7 | 8 | 7
Gait disturbance (General disorders) | 0 | 0 | 1 | 0
Hyperplasia (General disorders) | 0 | 0 | 0 | 1
Induration (General disorders) | 1 | 0 | 1 | 1
Influenza like illness (General disorders) | 2 | 0 | 1 | 0
Irritability (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0
Medical device pain (General disorders) | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 1 | 0
Nodule (General disorders) | 1 | 0 | 1 | 2
Non-cardiac chest pain (General disorders) | 2 | 0 | 1 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 4 | 2 | 2 | 3
Pain (General disorders) | 1 | 1 | 1 | 2
Pyrexia (General disorders) | 1 | 0 | 3 | 1
Spinal pain (General disorders) | 1 | 0 | 0 | 1
Suprapubic pain (General disorders) | 1 | 0 | 0 | 0
Swelling (General disorders) | 0 | 0 | 0 | 1
Temperature intolerance (General disorders) | 2 | 0 | 0 | 0
Xerosis (General disorders) | 1 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 3 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 1 | 1 | 0 | 2
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 1 | 0 | 2
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 4 | 3
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0
Vulvitis (Infections and infestations) | 0 | 0 | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1
Incision site oedema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Scar (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 5 | 1 | 6 | 3
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 1 | 1
Amylase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 0 | 0
Bilirubin conjugated increased (Investigations) | 0 | 0 | 1 | 0
Blast cell count increased (Investigations) | 0 | 0 | 1 | 0
Blood albumin decreased (Investigations) | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 2 | 1
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 2 | 0 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 3 | 0 | 3 | 1
Blood lactate dehydrogenase decreased (Investigations) | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 2 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 1 | 0
Blood urea increased (Investigations) | 2 | 1 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 1
Carbon dioxide decreased (Investigations) | 0 | 0 | 2 | 1
Cardiac murmur (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 1 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 2 | 1 | 3
Glomerular filtration rate decreased (Investigations) | 1 | 0 | 1 | 1
Glomerular filtration rate increased (Investigations) | 0 | 1 | 0 | 0
Granulocyte count increased (Investigations) | 1 | 1 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1 | 0
Lymph node palpable (Investigations) | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 2 | 0 | 1
Mean cell haemoglobin concentration increased (Investigations) | 0 | 1 | 0 | 0
Mean cell volume increased (Investigations) | 0 | 0 | 1 | 0
Mean platelet volume decreased (Investigations) | 0 | 0 | 0 | 1
Metamyelocyte count increased (Investigations) | 0 | 0 | 1 | 0
Monocyte count increased (Investigations) | 1 | 0 | 1 | 0
Myelocyte count increased (Investigations) | 0 | 0 | 1 | 0
Promyelocyte count increased (Investigations) | 0 | 0 | 1 | 0
Protein total decreased (Investigations) | 0 | 1 | 0 | 0
Protein total increased (Investigations) | 0 | 0 | 0 | 1
Protein urine present (Investigations) | 0 | 1 | 0 | 0
Red cell distribution width increased (Investigations) | 0 | 0 | 1 | 0
Specific gravity urine decreased (Investigations) | 1 | 0 | 0 | 1
Specific gravity urine increased (Investigations) | 0 | 1 | 1 | 1
Urine ketone body present (Investigations) | 1 | 0 | 1 | 0
Urine leukocyte esterase positive (Investigations) | 0 | 0 | 1 | 0
Urine output increased (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 5 | 2 | 2 | 3
Weight increased (Investigations) | 0 | 0 | 0 | 1
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 4 | 4 | 6
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2
Zinc deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 5 | 9 | 9
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1
Lower extremity mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 6 | 3 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Upper extremity mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Acanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1 | 2
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2 | 2 | 4
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 4 | 3
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Warty dyskeratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Coordination abnormal (Nervous system disorders) | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 3 | 2
Dysguesia (Nervous system disorders) | 1 | 3 | 3 | 1
Headache (Nervous system disorders) | 1 | 4 | 1 | 6
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 1 | 1
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 1 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
VII nerve paralysis (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 2 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 2 | 0 | 1
Illusion (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 3 | 0
Libido decreased (Psychiatric disorders) | 0 | 2 | 0 | 0
Mood altered (Psychiatric disorders) | 1 | 0 | 0 | 0
Self-induced vomiting (Psychiatric disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 1
Urinary tract disorder (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urine flow decreased (Renal and urinary disorders) | 1 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Nipple pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 3 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 3 | 1 | 5 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 3 | 2 | 4
Blister (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 4
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 4 | 4 | 3 | 3
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 4 | 2 | 6 | 5
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 2
Lentigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Leukoplakia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Milia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0
Papule (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0
Parakeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Perivascular dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 5 | 3 | 5 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 7 | 5 | 6
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Sebaceous gland disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 3 | 3 | 3
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 4 | 1 | 3
Skin plaque (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Sinus operation (Surgical and medical procedures) | 0 | 1 | 0 | 0
Extremity necrosis (Vascular disorders) | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 1 | 1 | 2
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 2
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.